CLINICAL TRIAL: NCT00496795
Title: Molecular Markers Predictive Response to Dose Dense Chemotherapy With Epirubicin and Docetaxel in Sequences for Locally Advanced Breast Cancer.
Brief Title: Predictors for Response to Dose-dense Docetaxel and Epirubicin Breast Cancer
Acronym: DDP
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Hans Petter Eikesdal, Professor, University of Bergen
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Ethics committee 079.06; NSD 14918; 14918 (Other: Helse Vest IKT)
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Stage III Breast Cancer AJCC V7
Keywords: Breast cancer, chemoresistance, predictive markers.
MeSH Terms: conditions — Breast Neoplasms | interventions — Epirubicin

STUDY DESIGN:
Intervention Model Description: Sequential epirubicin and docetaxel
Oversight: Data Monitoring Committee: No

ARMS (1):
- epirubicin/docetaxel sequential (Other): Epirubicin/docetaxel sequential, i.e. one arm study with Epirubicin 4 cycles 60 mg/m2 q2w, followed by docetaxel 4 cycles, 100 mg/m2 q2w. Each course with pegfilgrastim.
  Interventions: Other: epirubicin/docetaxel sequential

INTERVENTIONS:
Other: epirubicin/docetaxel sequential — Epirubicin 60 mg/m2, q2w 4 cycles. Followed by docetaxel 100 mg/m2 q2w 4 cycles
  Other Names: Farmorubicin (Pfizer)

SUMMARY:
Molecular markers predicting response to dose dense chemotherapy with epirubicin and docetaxel in sequence for locally advanced breast cancer

Protocol summary.

Principal Investigator Hans P. Eikesdal, Professor, Dept. of Oncology, Haukeland University Hospital & Dept. of Clinical Science, University of Bergen

Project leader: Professor Per Eystein Lønning, Dept. of Oncology, Haukeland University Hospital & Dept. of Clinical Science, University of Bergen

Collaborators. Dept of Surgery - Responsible: Turid Aas, Consultant Surgeon

Participants. Dept of Oncology Stephanie Geisler, Consultant Oncologist Jurgen Geisler, Consultant Oncologist

Type of Study Phase II, Translational research

Scientific aims: Addressing factors predicting response to dose intensive epirubicin followed by docetaxel sequential therapy

Treatment regimen: epirubicin 60 mg/m2 on a 2 weekly basis x 4 followed by docetaxel 100 mg/m2 2-weekly x 4.

Patients: Breast cancer patients below 65 years of age suffering from large (>4 cm largest diameter, non-inflammatory and / or N2-N3) primary breast cancer.

.

Clinical aim: Assessing responsiveness to this dose intensive regimen.

Number of patients to be enrolled: 60 - 100

DETAILED DESCRIPTION:
Aim The scientific aim of this study is to explore mechanisms of resistance to chemotherapy in breast cancer. To do so, we explore molecular parameters predicting response to chemotherapy administered prior to local therapy in large, primary breast cancers.

Background Neoadjuvant (primary medical) therapy has got wide acceptance as primary therapy in breast cancer. In addition, this treatment provides an optimal setting studying the mechanisms of drug resistance in human cancers.

Considering chemotherapy for primary breast cancer treatment, contemporary trend has been to treat these tumors more aggressively. High-dose therapy involving stem cell support is not advocated, as this has not been shown to improve long-term survival in early breast cancer. However, the attitude in general has been toward a more aggressive approach within the frame of "conventional" therapy.

Based on theoretical modeling, an alternative approach, "dose-dense" therapy, has been advocated. Recently, that concept was brought to the test in two adjuvant trials. Thus, Citron et al applying doxorubicin, paclitaxel and cyclofosfamide revealed an improved outcome for dose-dense (2-weekly) administration compared to regular 3-weekly scheduling. In contrast, the German GEPARDUO study reported doxorubicin plus cyclophosphamide and docetaxel, given in sequence on a 3-weekly basis (8 cycles), to be superior to doxorubicin and docetaxel given in concert on a 2-weekly basis for 4 cycles. However, the doses administered (doxorubicin 50 versus 60 mg/m2; docetaxel 75 versus 100 mg/m2) was unequal, meaning total drug dose exposure differed between the two treatment arms. While more data are warranted, a reasonable interpretation of available data suggest sequential administration of different compounds in a dose-density approach to be a suitable regimen provided adequate total doses are given.

Rationale for regimen Considering anthracyclines, most regimens today combine either epirubicin or doxorubicin in concert with 5-fluorouracil and cyclophosphamide. However, based on the evidence in the literature, it is not clear what the contribution of 5-FU or cyclophosphamide is to the effectiveness of such regimens, in particular not when a taxane is administered in sequence or concert. Thus, the NSABP-group has abandoned use of 5-FU from their adjuvant regimen. Considering cyclophosphamide, this compound seems to add to the carcinogenetic effect of anthracyclines enhancing the risk of secondary leukemia, while the contribution to the antitumor efficacy of the regimen remains uncertain. The taxanes are known to have significant antitumor effects in breast cancer when administered as monotherapy. Considering docetaxel, the dose generally advocated for monotherapy is 100 mg/m2, while a dose of 75mg/m2 is recommended for combined use. Thus, the potential exists that the dose for combined use may be sub-optimal in some patients.

Justification for a sequential approach is further supported by studies in metastatic breast cancer.

Scientific aims While many mechanisms of resistance have been identified in experimental systems, we have little knowledge what may be the cause of drug resistance in human cancers. The factors so far identified that have been found associated with resistance to chemotherapy in breast cancer are amplification of HER-2 / Topo-II and mutations affecting TP53.

Recently, several groups have explored responsiveness to chemotherapy using mRNA microarrays. While these studies consistently identified different gene profiles correlating to responsiveness to different regimens, the predictive value was too low for clinical application. Moreover, the results did not add to our understanding of the biological mechanisms causing drug resistance. In contrast, studies exploring different forms of cancer have started to reveal specific gene alterations, in particular affecting pathways of DNA damage repair or apoptosis in relation to drug resistance. Thus, our primary aim is to explore potential gene disturbances based on functional hypotheses.

A major issue identifying mechanisms of drug resistance is to explore different compounds on a monodrug basis. Clinically, the major reason for combining or administering sequentially an anthracycline and a taxane is the efficacy of each compound combined with a significant lack of cross-resistance. Administered as a combined schedule, this limits the possibility of identifying the mechanisms of resistance / sensitivity to each compound individually. Provided that a sequential regimen provides the same efficacy as a combined schedule, such an approach is justified ethically. Thus, for a patient given 2 and 3 drugs in concert, the potential may be they respond to one drug only, while having the toxicity of the other compounds. In case of non-responsiveness to a single compound, this may be exchanged for an alternative treatment option. This contrasts the possibilities provided in the adjuvant setting. In adjuvant therapy, there is no way by which we may assess the response to individual drugs; thus the different compounds have to administer in concert.

Based on what is said above, we consider sequential dose-dense treatment using epirubicin and docetaxel sequentially to be a feasible treatment option.

Treatment regimen Each patient will receive 4 cycles of epirubicin 60 mg/m2 given at 2 weekly intervals together with G-CSF. Thereafter, docetaxel 100 mg/ m2 will be given at 2 weekly intervals for 4 cycles. Patients revealing positivity for HER2 status will have trastuzumab (Herceptin) implemented together with docetaxel but not during anthracycline treatment.

Staging at baseline

After given informed consent, patients will be staged as follows:

* MRI of both breasts
* Chest X-ray
* Liver ultrasound (in case metastases are suspected or verified; to be followed by CT and / or MRI confirmation)
* Skeletal scintigram. Any positive findings to be confirmed by subsequent X-ray / CT and / or MRI
* ECG
* LVEF (Left Ventricular Ejection Fraction)

Response evaluation Response will be evaluated based on clinical examination and MRI, each assessment to be done separately.

Clinical examination will be performed prior to commencing therapy (before surgical biopsy) and subsequently at 4, 6 and 8 weeks on therapy. Response will be classified according to the common "RECIST" criteria. An important exception is to be made. As argued in a previous protocol, we consider the RECIST definition of "progressive disease" as a 20% increase in the sum of the largest tumor diameters to be too liberal with respect to large primary tumors. Based on experience in our clinic, we believe the definition of progressive disease as an increase of > 25% in the product of the largest tumor diameter and its perpendicular (the previous common UICC criteria) to be a more suitable definition, protecting patients from undergoing deterioration of their clinical condition. This is in accordance to our previous experience.

In case of "progressive disease" at any stage during epirubicin treatment, the patient will terminate epirubicin immediately and go ahead with docetaxel treatment. In case of progressive disease on docetaxel treatment, further therapy is left to the physician's discretion.

Considering MRI assessment, this should be performed prior to commencing therapy, in the interval following the 4th cycle of epirubicin (prior to commencing docetaxel) and after the 4th cycle of docetaxel, prior to surgery.

Tissue sampling

1. Each patient will undergo a surgical biopsy prior to commencing treatment.
2. A Tru-cut biopsy should be obtained 24 hours after administration of the first epirubicin cycle to assess "immediate" alterations in response to cytotoxic damage.
3. Immediately prior to commencing treatment with docetaxel, a third sample (this time a Tru-Cut biopsy) is obtained for snap-freezing.
4. A Tru-cut biopsy should be obtained 24 hours after administration of the first docetaxel cycle to assess "immediate" alterations in response to cytotoxic damage.
5. Finally, tumor tissue is collected and snap-frozen at surgery following docetaxel therapy.

Bone marrow aspiration A single unilateral bone marrow aspiration is performed prior to commencing chemotherapy treatment.

Study Endpoint

* Primary endpoint is to correlate molecular parameters to objective response to each of the 2 regimens applied.
* Secondary endpoint are

  : - to correlate molecular parameters to relapse-free and overall survival
* to identify and explore characteristics of epithelial and mesenchymal stem cells isolated in tumor tissue and bone marrow

Surgery While many centers practice breast conservative surgery for tumors successfully downstaged by primary medical treatment, in general we have applied a conservative approach, advocating mastectomy. However, downstaging for limited surgery is not a primary or secondary endpoint of this study. In general, we will advocate mastectomy also for patients with a clinical complete response. However, this practice may change based on contemporary results from other centers, and the protocol allow limited surgery at the physicians discretion in individual patients.

Laboratory Investigations The area of molecular biology is rapidly developing with respect to biological knowledge as well as technical analytical methods. Thus, it is not possible to predict upfront which genes may be of particular interest in 5 years from know; neither is it possible to foresee completely which laboratory methods will be available. Our aim is to explore potential genetic alterations explaining the mechanisms of drug resistance. While it is not possible to predict in detail, the aim of the study and all analysis to be conducted should aim at this major goal.

Number of patients to be enrolled The study is an exploratory translational study. Thus, we do not know the number of patients expected to achieve a clinical or pathological complete response. Currently, on average 20 patients are referred to our Department for a diagnosis of locally advanced breast cancer on an annual basis; including patients with tumors measuring between 4 and 5 cm in diameter, we estimate the total number may be somewhere between 30 and 40 patients per year. From this cohort, we estimate an average number of 20 patients to be enrolled in the study on an annual basis. Our aim is to recruit 100 patients with a minimum of 60.

Publication Our aim is to publish the results from this study in peer-reviewed international journals with contributors from the clinic and laboratory as authors.

References; from the Trial Administrator upon request.

ELIGIBILITY:
Inclusion Criteria:

* Primary breast cancer >4cm in diameter and / or lymph node status N2-3.
* Age 65 years or younger
* "Limited" distant metastases allowed, but patients with massive distant metastases should be excluded
* Willing to participate in the study

Exclusion Criteria:

* Known allergy toward any of the cytotoxic compounds to be administered (epirubicin and doxorubicin)
* Liver enzymes > 2 times upper normal limit or bilirubin > 3 times upper normal limit
* Other medical conditions making them unfit for dose-dense therapy
* Cardiac insufficiency; for patients not to receive trastuzumab, decision whether to exclude such patients will be at the physicians discretion. Considering patients with HER-2 positive tumors who should have trastuzumab, exclusion criteria will be according to the NBCG (Norwegian Breast Cancer Group) general guidelines (www.NBCG.net).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-09; Primary Completion 2016-05 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
To correlate molecular parameters to objective response to each of the 2 regimens applied. | 10 years
  To correlate molecular parameters to objective response to sequential dose-dense therapy with epirubicin followed by docetaxel in primary locally advanced breast cancer.

SECONDARY OUTCOMES:
To correlate molecular parameters to relapse-free and overall survival. | 10 years
To identify and explore characteristics of epithelial and mesenchymal stem cells isolated in tumor tissue and bone marrow | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Per E Lonning, MD PhD, Study Chair — Section of Oncology, Institute of Medicine, University of Bergen, Haukeland University Hospital
Locations (1):
- Dept of Oncology, Bergen, Norway

REFERENCES:
- [Derived] Hatletvedt ND, Engebrethsen C, Geisler J, Geisler S, Aas T, Lonning PE, Gansmo LB, Knappskog S. The impact of functional MDM2-polymorphisms on neutrophil counts in breast cancer patients during neoadjuvant chemotherapy. BMC Cancer. 2025 Feb 20;25(1):308. doi: 10.1186/s12885-025-13675-2. PMID 39979836
- [Derived] Venizelos A, Engebrethsen C, Deng W, Geisler J, Geisler S, Iversen GT, Aas T, Aase HS, Seyedzadeh M, Steinskog ES, Myklebost O, Nakken S, Vodak D, Hovig E, Meza-Zepeda LA, Lonning PE, Knappskog S, Eikesdal HP. Clonal evolution in primary breast cancers under sequential epirubicin and docetaxel monotherapy. Genome Med. 2022 Aug 11;14(1):86. doi: 10.1186/s13073-022-01090-2. PMID 35948919

DOCUMENTS (2):
  • Study Protocol (2006-03-16): https://cdn.clinicaltrials.gov/large-docs/95/NCT00496795/Prot_000.pdf
  • Informed Consent Form (2006-08-23): https://cdn.clinicaltrials.gov/large-docs/95/NCT00496795/ICF_001.pdf